CLINICAL TRIAL: NCT06301321
Title: The Evaluation and Comparison of BCR-ABL p210 mRNA Transcripts (%IS Unit) Results Between Dr. PCR™ BCR-ABL1 Major IS Detection Kit (Optolane) and QXDx™ BCR-ABL %IS Kit (Bio-Rad) in Chronic Myeloid Leukemia Patients
Acronym: BCR-ABL1
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Weerapat Owattanapanich, Associate professor, Siriraj Hospital
Other Study IDs: 461_2566
Record Dates: First submitted 2024-02-20; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: BCR-ABL p210 mRNA transcripts; Dr. PCR™ BCR-ABL1 Major IS Detection; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, there are many commercial kits for detecting BCR-ABL fusion transcripts. The QXDx™ BCR-ABL %IS kit (Bio-Rad, Hercules, CA, USA) is the first ddPCR-based in vitro diagnostics (IVD) product with the US Food and Drug Administration clearance and European Conformity (CE) mark which launched in 2017. Dr. PCR™ BCR-ABL1 Major IS Detection Kit (Optolane, South Korea) is one of CE-IVD commercial kits based on digital RT-PCR. Both commercial kits are digital PCR-based, also evaluated their correlation, pros and cons in order for users to select a reagents kit that are appropriate for themselves.

DETAILED DESCRIPTION:
Today, there are many commercial kits for detecting BCR-ABL fusion transcripts. The QXDx™ BCR-ABL %IS kit (Bio-Rad, Hercules, CA, USA) is the first ddPCR-based in vitro diagnostics (IVD) product with the US Food and Drug Administration clearance and European Conformity (CE) mark which launched in 2017. Dr. PCR™ BCR-ABL1 Major IS Detection Kit (Optolane, South Korea) is one of CE-IVD commercial kits based on digital RT-PCR. Both commercial kits are digital PCR-based, also evaluated their correlation, pros and cons in order for users to select a reagents kit that are appropriate for themselves.

Objectives 1.To evaluate and comparison of BCR-ABL p210 mRNA transcripts (%IS unit) results from two detection kit ; Dr. PCR™ BCR-ABL1 Major IS Detection Kit (Optolane) VS QXDx™ BCR-ABL %IS Kit (Bio-Rad) in chronic myeloid leukemia (CML) patients Secondary objective 2.To be used as a standard inspection method of the Hematology laboratory at Siriraj Hospital Inclusion criteria

1. Leftover RNA samples from CML patients were recruited from the Hematology Laboratory Division of Hematology Department of Medicine Faculty of Medicine, Siriraj Hospital Mahidol University, after TKI treatment and regular follow-ups or newly diagnosed.
2. All samples were successively tested by QXDx™ BCR-ABL %IS Kit (Bio-Rad) which used Droplet Digital PCR (ddPCR) technique.

Exclusion criteria

1.In adequate or poor-quality specimen

ELIGIBILITY:
Inclusion Criteria:

* Leftover RNA samples from CML patients were recruited from the Hematology Laboratory Division of Hematology Department of Medicine Faculty of Medicine, Siriraj Hospital Mahidol University, after TKI treatment and regular follow-ups or newly diagnosed.
* All samples were successively tested by QXDx BCR-ABL %IS Kit (Bio-Rad) which used Droplet Digital PCR (ddPCR) technique.

Exclusion Criteria:

* In adequate or poor-quality specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients 18 years and older who were newly diagnosis and known to have CML
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  Positive predictive value, negative predictive value and AUC. A p-value < 0.05 was considered statistically significant difference.
Specificity | Through study completion, an average of 1 year
  Positive predictive value, negative predictive value and AUC. A p-value < 0.05 was considered statistically significant difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol